CLINICAL TRIAL: NCT07235826
Title: Evaluation of the Efficacy of Streptococcus Salivarius Evol12® in the Reduction of Recurrent Adenotonsillitis in Children: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Cross-over Clinical Trial
Brief Title: Evaluation of the Efficacy of Streptococcus Salivarius Evol12® in the Reduction of Recurrent Adenotonsillitis in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 140_16luglio_BactoblisEvol
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Tonsillitis
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either Streptococcus salivarius Evol12® (Bactoblis® Evol) for 3 months followed by placebo for 3 months, or the reverse sequence, with a 7-day wash-out period between treatment phases.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design: participants, caregivers, investigators, and outcome assessors are blinded to treatment allocation. The probiotic and placebo tablets are identical in appearance, packaging, and labeling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bactoblis® Evol (Experimental): Participants randomized to Sequence A will receive Streptococcus salivarius Evol12® (Bactoblis® Evol) for 3 months, followed by a 7-day wash-out, then matching placebo for 3 months. Bactoblis® Evol is taken as 1 orodispersible tablet nightly, allowed to dissolve slowly in the mouth.
  Interventions: Dietary Supplement: Bactoblis® Evol (Streptococcus salivarius Evol12®)
- Placebo (Placebo Comparator): Participants randomized to Sequence B will receive matching placebo for 3 months, followed by a 7-day wash-out, then Streptococcus salivarius Evol12® (Bactoblis® Evol) for 3 months. The placebo tablets are identical in appearance, taste, and packaging to the active product.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bactoblis® Evol (Streptococcus salivarius Evol12®) — Bactoblis® Evol is an orodispersible tablet containing the probiotic strain Streptococcus salivarius Evol12® (LMG P-33696), used to support the balance of the oral microbiota. Each tablet is taken once daily in the evening, allowing it to dissolve slowly in the mouth without chewing, eating, or drinking afterward. Treatment is administered for 3 consecutive months during each treatment period. The product is manufactured by PharmExtracta S.p.A., Pontenure, Italy.
  Arms: Bactoblis® Evol
Other: Placebo — Matching placebo orodispersible tablet identical in appearance, flavor, and packaging to Bactoblis® Evol but without the active probiotic strain. Administered once daily in the evening for 3 months during the assigned treatment period.
  Other Names: Placebo (matching orodispersible tablet)
  Arms: Placebo

SUMMARY:
This prospective, multicenter, randomized, double-blind, placebo-controlled, cross-over clinical trial will evaluate the efficacy and safety of Streptococcus salivarius Evol12® (Bactoblis® Evol) in reducing the recurrence and duration of acute febrile adenotonsillitis in children aged 3 to 11 years. Participants will receive either the probiotic or a matching placebo for 3 months, followed by a 7-day wash-out and a second 3-month treatment period with the alternative product. The study will assess changes in the incidence and duration of adenotonsillar episodes, antibiotic use, school absences, and sleep quality.

DETAILED DESCRIPTION:
Recurrent adenotonsillitis in children is a frequent and burdensome condition, often leading to repeated antibiotic use, missed school days, and sleep disturbances. Streptococcus salivarius is a naturally occurring commensal bacterium of the oral microbiota with demonstrated ability to inhibit Streptococcus pyogenes and other pathogens responsible for pharyngotonsillitis. Streptococcus salivarius Evol12® is a novel probiotic strain with a safe microbiological profile and no antibiotic resistance, developed to restore oral microbial balance and reduce recurrent infections of the upper airways.

This non-profit, prospective, multicenter, randomized, double-blind, placebo-controlled, cross-over study will enroll 200 pediatric participants aged 3 to 11 years with a history of at least three documented episodes of acute febrile adenotonsillitis in the preceding 12 months. Participants will be randomized to receive either one orodispersible tablet of S. salivarius Evol12® (Bactoblis® Evol, PharmExtracta S.p.A., Italy) daily in the evening for 3 months followed by placebo for 3 months, or vice versa, with a 7-day wash-out period between treatments.

The primary objective is to evaluate the efficacy of S. salivarius Evol12® in reducing the duration and recurrence of acute febrile adenotonsillitis, as measured by the Wisconsin Upper Respiratory Symptom Survey for Kids (WURSS-K).

Secondary objectives include assessment of sleep disorders (OSA-18 questionnaire), number and duration of feverish episodes, school days missed, antibiotic use, and symptom severity (e.g., sore throat, tonsil exudate, difficulty swallowing, otitis, cough, and fatigue).

Ethical approval has been granted by the Ethics Committee of the University of Urbino Carlo Bo (Minutes No. 96, July 24, 2025).

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 3 to 11 years.
* History of ≥3 documented episodes of acute adenotonsillitis within the previous 12 months, each characterized by fever ≥38°C.
* Signed and accepted informed consent from a parent or legal guardian.

Exclusion Criteria:

* Total obstruction of the nasal cavities.
* Uncontrolled gastroesophageal reflux disease.
* Unilateral tonsillar enlargement.
* Previous tonsil reduction surgery.
* Lack of parental or legal guardian consent to participate in the study.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in recurrence of acute febrile adenotonsillitis | 6 months
  Number of febrile adenotonsillitis episodes occurring during the 6-month study period. Outcomes will be assessed using the Wisconsin Upper Respiratory Symptom Survey for Kids (WURSS-K), completed during each febrile episode to record symptom severity and quality of life.
Reduction in duration of acute febrile adenotonsillitis episodes | 6 months
  Duration (in days) of each febrile adenotonsillitis episode during the 6-month study period, assessed using the Wisconsin Upper Respiratory Symptom Survey for Kids (WURSS-K) completed by caregivers during illness episodes.

SECONDARY OUTCOMES:
Occurrence of adenotonsillar symptoms | 6 months
  Number of adenotonsillar symptom episodes (fever ≥38°C, sore throat, tonsil exudate, difficulty swallowing, earache, acute otitis media, fatigue or joint pain, swollen lymph nodes, or cough) reported by parents or guardians using an episode symptom card.
Duration of adenotonsillar symptoms | 6 months
  Total duration (in days) of adenotonsillar symptom episodes (fever ≥38°C, sore throat, tonsil exudate, difficulty swallowing, earache, acute otitis media, fatigue or joint pain, swollen lymph nodes, or cough) reported by parents or guardians using an episode symptom card.
Change in sleep-related quality of life assessed by the Obstructive Sleep Apnea-18 (OSA-18) questionnaire | 6 months
  Assessment of changes in sleep-related quality of life using the Obstructive Sleep Apnea-18 (OSA-18) questionnaire completed by the parent or legal guardian.
  The OSA-18 total score ranges from 18 to 126, with higher scores indicating a worse sleep-related quality of life. The questionnaire evaluates symptoms and impact across five domains: sleep disturbance, physical suffering, emotional distress, daytime problems, and caregiver concerns.
Number of school days missed | 6 months
  Total number of school days missed due to adenotonsillar infections during the study period, as recorded in the daily symptom card.
Number of antibiotic treatments prescribed for adenotonsillar infections | 6 months
  otal number of antibiotic treatment courses prescribed for adenotonsillar infections during the 6-month study period, as reported by parents or legal guardians on the episode symptom card.
Duration of antibiotic treatment for adenotonsillar infections | 6 months
  Total duration (in days) of antibiotic treatment courses prescribed for adenotonsillar infections during the 6-month study period, as reported by parents or legal guardians on the episode symptom card.

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Urbino Carlo Bo, Urbino, PU (Pesaro E Urbino), Italy

REFERENCES:
- [Background] Di Pierro F, Thacharodi A, Kumaraswami M, Bertuccioli A, Tanda ML, Zerbinati N. Description of the draft genome sequence of Streptococcus salivarius eK12, a derivative of the probiotic strain Streptococcus salivarius K12 with a modified plasmid. Microbiol Resour Announc. 2025 Aug 14;14(8):e0035525. doi: 10.1128/mra.00355-25. Epub 2025 Jul 8. PMID 40626761
- [Background] Bertuccioli A, Cardinali M, Micucci M, Rocchi MBL, Palazzi CM, Zonzini GB, Annibalini G, Belli A, Sisti D. Efficacy of Streptococcus salivarius Blis K12 in the Prevention of Upper Respiratory Tract Infections in Physically Active Individuals: A Randomized Controlled Trial. Microorganisms. 2024 Oct 26;12(11):2164. doi: 10.3390/microorganisms12112164. PMID 39597553
- [Background] Di Pierro F, Colombo M, Zanvit A, Rottoli AS. Positive clinical outcomes derived from using Streptococcus salivarius K12 to prevent streptococcal pharyngotonsillitis in children: a pilot investigation. Drug Healthc Patient Saf. 2016 Nov 21;8:77-81. doi: 10.2147/DHPS.S117214. eCollection 2016. PMID 27920580
- [Background] La Torre F, Sota J, Insalaco A, Conti G, Del Giudice E, Lubrano R, Breda L, Maggio MC, Civino A, Mastrorilli V, Loconte R, Natale MF, Celani C, Romeo M, Patroniti S, Gentile C, Vitale A, Caggiano V, Gaggiano C, Diomeda F, Cattalini M, Lopalco G, Emmi G, Parronchi P, Gentileschi S, Cardinale F, Aragona E, Shahram F, Marino A, Barone P, Moscheo C, Ozkiziltas B, Carubbi F, Alahmed O, Iezzi L, Ogunjimi B, Mauro A, Tarsia M, Mahmoud AAA, Giardini HAM, Sfikakis PP, Laskari K, Wiesik-Szewczyk E, Hernandez-Rodriguez J, Frediani B, Gomez-Caverzaschi V, Tufan A, Almaghlouth IA, Balistreri A, Ragab G, Fabiani C, Cantarini L, Rigante D. Preliminary data revealing efficacy of Streptococcus salivarius K12 (SSK12) in Periodic Fever, Aphthous stomatitis, Pharyngitis, and cervical Adenitis (PFAPA) syndrome: A multicenter study from the AIDA Network PFAPA syndrome registry. Front Med (Lausanne). 2023 Feb 16;10:1105605. doi: 10.3389/fmed.2023.1105605. eCollection 2023. PMID 36873863
- [Background] Wescombe PA, Hale JD, Heng NC, Tagg JR. Developing oral probiotics from Streptococcus salivarius. Future Microbiol. 2012 Dec;7(12):1355-71. doi: 10.2217/fmb.12.113. PMID 23231486
- [Background] Rajasekaran JJ, Krishnamurthy HK, Bosco J, Jayaraman V, Krishna K, Wang T, Bei K. Oral Microbiome: A Review of Its Impact on Oral and Systemic Health. Microorganisms. 2024 Aug 29;12(9):1797. doi: 10.3390/microorganisms12091797. PMID 39338471